CLINICAL TRIAL: NCT06883305
Title: A Randomised, Double-blind, Placebo-controlled, Parallel Group, Multicentre, Phase III Study to Evaluate the Efficacy and Safety of Tezepelumab in Adult Participants With Moderate to Very Severe Chronic Obstructive Pulmonary Disease
Brief Title: A Study to Investigate the Efficacy and Safety of Tezepelumab in Adult Participants With Moderate to Very Severe COPD (D5241C00006)
Acronym: EMBARK
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5241C00006
Record Dates: First submitted 2025-03-03; First posted 2025-03-19 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Moderate COPD; Severe COPD; Very Severe COPD; chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — tezepelumab

STUDY DESIGN:
Intervention Model Description: Participants will be randomised in a ratio of 1:1:1 to receive Dose 1 of tezepelumab, Dose 2 of tezepelumab or matching placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose 1 of Tezepelumab (Experimental): Tezepelumab, SC, Q4W
  Interventions: Biological: Tezepelumab
- Dose 2 of Tezepelumab (Experimental): Tezepelumab, SC, Q4W
  Interventions: Biological: Tezepelumab
- Matching Placebo (Placebo Comparator): Matching placebo, SC, Q4W
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Tezepelumab — Tezepelumab subcutaneous injection
  Arms: Dose 1 of Tezepelumab; Dose 2 of Tezepelumab
Other: Placebo — Placebo subcutaneous injection
  Arms: Matching Placebo

SUMMARY:
A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel Group, Phase 3 Study to Evaluate the Efficacy and Safety of Tezepelumab in Adults with Moderate to Very Severe Chronic Obstructive Pulmonary Disease (COPD)

DETAILED DESCRIPTION:
This is a Phase 3, multicenter, randomized, double-blind, placebo-controlled, parallel group study to evaluate the safety and efficacy of tezepelumab in adults with moderate to very severe chronic obstructive pulmonary disease (COPD) receiving inhaled maintenance therapy and having had at least 2 moderate, or 1 severe, COPD exacerbations in the 12 months prior to Visit 1. Subjects will receive monthly subcutaneous injection of one of two different doses of tezepelumab, or placebo, with a maximum treatment duration of 76 weeks and a minimum of 52 weeks. The study also includes a off-treatment safety follow-up period of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. ≥40 to ≤80 years old
2. COPD diagnosis ≥1 year,
3. Post-BD FEV1 ≥ 20% and ≤ 70% PN, FEV1/FVC <0.70 at screening
4. Triple (ICS+LABA+LAMA) or dual inhaled COPD therapy, if triple therapy is considered not appropriate, ≥3 consecutive months prior to V1
5. ≥2 moderate or ≥1 severe COPD exacerbations in the prior year; At least 1 of 2 moderate exacerbations must require the use of systemic corticosteroids. At least one of the previous exacerbations should be confirmed to have occurred while the participant was on triple or dual inhaled maintenance therapy
6. EOS ≥ 150 cells/μL during screening
7. CAT ≥15 at screening
8. Former or current smokers ≥10 pack-years

Exclusion Criteria:

1. Clin. important pulmonary disease or radiological findings suggestive of a respiratory disease other than COPD
2. Asthma, incl. pediatric, or ACOS
3. Any unstable disorder that can impact participants safety or study outcomes
4. Tuberculosis requiring treatment within 12 months prior V2
5. Malignancies current or past

   Concomitant therapies:
   * Macrolides (less than 6 months)
   * Systemic immuno-suppressive, -modulating medications
6. LTOT >4.0 L/min or O2 saturation <89% despite LTOT

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 990 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2029-03-13 (Estimated); Study Completion 2029-06-05 (Estimated)

PRIMARY OUTCOMES:
Annualised rate of moderate or severe COPD exacerbations | Baseline up to 76 weeks
  The annualised moderate or severe COPD exacerbation rate (based on exacerbations reported by the investigator) up to 76 weeks treatment period compared to placebo.

SECONDARY OUTCOMES:
Change from baseline in post-BD FEV1 | From baseline to Week 52
  Change from baseline in post-BD FEV1 at Week 52 compared to placebo. FEV1 is defined as the volume of air exhaled from the lungs in the first second of a forced expiration
Change from baseline in pre-dose/pre-bronchodilator (pre-BD) forced expiratory volume in 1 second (FEV1) | From baseline to Week 52
  Change from baseline in pre-BD FEV1 at Week 52 compared to placebo. FEV1 is defined as the volume of air exhaled from the lungs in the first second of a forced expiration.
Change from baseline in the St. George's Respiratory Questionnaire (SGRQ) total score | From baseline over 52 weeks
  Change from baseline in the SGRQ total score over 52 weeks compared to placebo.
  SGRQ is a disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease. Scores range from 0 to 100, with lower scores indicating better health status.
Annualised rate of moderate or severe COPD exacerbations among participants with EOS ≥ 300 cells/µL collected during screening visit. | Baseline up to 76 weeks
  The annualised moderate or severe COPD exacerbation rate (based on exacerbations reported by the investigator) up to 76 weeks treatment period compared to placebo among participants with EOS ≥ 300 cells/µL collected during screening visit.
Annualised rate of severe COPD exacerbations | Baseline up to 76 weeks
  The annualised severe COPD exacerbation rate (based on exacerbations reported by the investigator) up to 76 weeks treatment period compared to placebo.
Annualised rate of COPD exacerbations requiring ER visit and/or hospitalisation | Baseline up to 76 Weeks
  The annualised rate of COPD exacerbation requiring ER visit and/or hospitalisation up to 76 weeks treatment period compared to placebo.
Clinical meaningful improvement in St. George's Respiratory Questionnaire (SGRQ) total score | From baseline over 52 weeks
  Participants achieving a clinically meaningful improvement from baseline in SGRQ total score (4-point score decrease) over 52 weeks.
  SGRQ is a disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease. Scores range from 0 to 100, with lower scores indicating better health status.
Change from baseline in the COPD assessment Test (CAT) total score | From baseline over 52 weeks
  Change from baseline in the CAT total score over 52 weeks
  CAT is an 8-item PRO that measures the impact of COPD on the health status of patients with COPD. The CAT has a scoring range of 0-40 with higher scores indicative of greater COPD impact on health status.
Clinical meaningful improvement in COPD Assessment Test (CAT) total score | From baseline over 52 weeks
  Participants achieving a clinically meaningful improvement from baseline in CAT total score (2-point score decrease) over 52 weeks.
  CAT is an 8-item PRO that measures the impact of COPD on the health status of patients with COPD. The CAT has a scoring range of 0-40 with higher scores indicative of greater COPD impact on health status.
Time to first moderate or severe COPD exacerbation | Baseline up to 76 weeks
  Time to first occurrence of moderate or severe COPD exacerbation up to 76 weeks.
Time to first severe COPD exacerbation | Baseline up to 76 weeks
  Time to first occurrence of severe COPD exacerbation up to 76 weeks.
Pharmacokinetics (PK): Serum trough concentrations | Baseline, Week 24, Week 36, Week 52
  Serum trough concentrations
Immunogenicity of anti-drug antibodies (ADA) | Baseline, Week 24, Week 36, Week 52
  Incidence of anti-drug antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Dave Singh, MD, Principal Investigator — Division of Infection, Immunity & Resp Medicine, The University of Manchester, United Kingdom
Locations (248):
- United States (59):
  - Research Site, Foley, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Sheffield, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Garden Grove, California
  - Research Site, Newport Beach, California
  - Research Site, Torrance, California
  - Research Site, Clearwater, Florida
  - Research Site, Cutler Bay, Florida
  - Research Site, DeBary, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Homestead, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Lithonia, Georgia
  - Research Site, Rincon, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Palos Hills, Illinois
  - Research Site, Winfield, Illinois
  - Research Site, Munster, Indiana
  - Research Site, Baltimore, Maryland
  - Research Site, Columbia, Maryland
  - Research Site, North Dartmouth, Massachusetts
  - Research Site, Farmington Hills, Michigan
  - Research Site, Saint Cloud, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Missoula, Montana
  - Research Site, Papillion, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, Sewell, New Jersey
  - Research Site, Toms River, New Jersey
  - Research Site, Buffalo, New York
  - Research Site, Cortland, New York
  - Research Site, Horseheads, New York
  - Research Site, High Point, North Carolina
  - Research Site, Kings Mountain, North Carolina
  - Research Site, New Bern, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Columbus, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, DuBois, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Rock Hill, South Carolina
  - Research Site, Franklin, Tennessee
  - Research Site, Johnson City, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, Humble, Texas
  - Research Site, Kerrville, Texas
  - Research Site, Mansfield, Texas
  - Research Site, Clearfield, Utah
  - Research Site, Morgantown, West Virginia
  - Research Site, Cudahy, Wisconsin
  - Research Site, Milwaukee, Wisconsin
- Brazil (11):
  - Research Site, Bragança Paulista
  - Research Site, Brasília
  - Research Site, Campinas
  - Research Site, Chapecó
  - Research Site, Curitiba
  - Research Site, Jaú
  - Research Site, Mossoró
  - Research Site, Porto Alegre
  - Research Site, Salvador
  - Research Site, São José do Rio Preto
  - Research Site, Vitória
- Canada (14):
  - Research Site, Calgary, Alberta
  - Research Site, Vancouver, British Columbia
  - Research Site, Ajax, Ontario
  - Research Site, Burlington, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Winchester, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint-Charles-Borromée, Quebec
  - Research Site, Saint-Laurent, Quebec
  - Research Site, Trois-Rivières, Quebec
  - Research Site, Saskatoon, Saskatchewan
- Chile (5):
  - Research Site, Concepción
  - Research Site, Curicó
  - Research Site, Quillota
  - Research Site, Santiago
  - Research Site, Talca
- China (44):
  - Research Site, Anyang
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Haikou
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Hengyang
  - Research Site, Heze
  - Research Site, Hohhot
  - Research Site, Huizhou
  - Research Site, Jinan
  - Research Site, Jinhua
  - Research Site, Linhai
  - Research Site, Loudi
  - Research Site, Nanchang
  - Research Site, Nanchong
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Pingxiang
  - Research Site, Qingdao
  - Research Site, Qingyuan
  - Research Site, Sanya
  - Research Site, Shanghai
  - Research Site, Shantou
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Shijiazhuang
  - Research Site, Suining Shi
  - Research Site, Taiyuan
  - Research Site, Taizhou
  - Research Site, Tianjin
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Xinxiang
  - Research Site, Xuzhou
  - Research Site, Yangzhou
  - Research Site, Yichang
  - Research Site, Yinchuan
  - Research Site, Zhangzhou
- Czechia (9):
  - Research Site, Brandýs nad Labem
  - Research Site, Brno
  - Research Site, Jindřichův Hradec
  - Research Site, Lovosice
  - Research Site, Ostrava
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Teplice
  - Research Site, Varnsdorf
- Research Site, København NV, Denmark
- Germany (9):
  - Research Site, Bendorf
  - Research Site, Berlin
  - Research Site, Haltern am See
  - Research Site, Hanover
  - Research Site, Immenhausen
  - Research Site, Lübeck
  - Research Site, Marburg
  - Research Site, Rosenheim
  - Research Site, Wiesbaden
- India (16):
  - Research Site, Ahmedabad
  - Research Site, Belagavi
  - Research Site, Coimbatore
  - Research Site, Dehradun
  - Research Site, Delhi
  - Research Site, Dwārka
  - Research Site, Faridabad
  - Research Site, Gūrgaon
  - Research Site, Kochi
  - Research Site, Kolkata
  - Research Site, Lucknow
  - Research Site, Madurai
  - Research Site, Mysuru
  - Research Site, Nagpur
  - Research Site, Pune
  - Research Site, Vadodara
- Italy (9):
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Montebelluna
  - Research Site, Napoli
  - Research Site, Pavia
  - Research Site, Roma
  - Research Site, Sassari
  - Research Site, Telese Terme
  - Research Site, Tradate
- Malaysia (7):
  - Research Site, Alor Star
  - Research Site, Kajang
  - Research Site, Kota Kinabalu
  - Research Site, Kuala Lumpur
  - Research Site, Kuala Terengganu
  - Research Site, Kuantan
  - Research Site, Kuching
- Mexico (13):
  - Research Site, Benito Juárez
  - Research Site, Chihuahua City
  - Research Site, Cuauhtémoc
  - Research Site, Cuernavaca
  - Research Site, Guadalajara
  - Research Site, Mérida
  - Research Site, Monterrey
  - Research Site, Morelia
  - Research Site, Oaxaca City
  - Research Site, San Juan del Río
  - Research Site, Tijuna
  - Research Site, Veracruz
  - Research Site, Zapopan
- Philippines (7):
  - Research Site, Iloilo City
  - Research Site, Las Piñas
  - Research Site, Manadaluyong City
  - Research Site, Manila
  - Research Site, Marilao
  - Research Site, Quezon City
  - Research Site, Tondo
- Poland (14):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Chrzanów
  - Research Site, Karczew
  - Research Site, Katowice
  - Research Site, Kielce
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Ostróda
  - Research Site, Piaseczno
  - Research Site, Poznan
  - Research Site, Pruszków
  - Research Site, Płock
- Slovakia (5):
  - Research Site, Humenné
  - Research Site, Košice
  - Research Site, Levice
  - Research Site, Martin
  - Research Site, Trnava
- South Korea (7):
  - Research Site, Anyang-si
  - Research Site, Daegu
  - Research Site, Iksan-si
  - Research Site, Jeonju
  - Research Site, Seoul
  - Research Site, Uijeongbu-si
  - Research Site, Wŏnju
- Spain (9):
  - Research Site, Barakaldo
  - Research Site, Barcelona
  - Research Site, Granada
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Palma de Mallorca
  - Research Site, Pamplona
  - Research Site, Seville
  - Research Site, Valencia
- United Kingdom (9):
  - Research Site, Bradford
  - Research Site, Brighton
  - Research Site, Cottingham
  - Research Site, Glasgow
  - Research Site, Halifax
  - Research Site, Leeds
  - Research Site, Portsmouth
  - Research Site, Tyne and Wear
  - Research Site, Wakefield

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/